CLINICAL TRIAL: NCT03785873
Title: A Single Arm Phase Ib/II Multi-Center Study of Nivolumab in Combination With Nanoliposomal-Irinotecan, 5-Fluorouracil, and Leucovorin as Second Line Therapy for Patients With Advanced Biliary Tract Cancer
Brief Title: Phase Ib/II Trial of Nal-Irinotecan and Nivolumab as Second-Line Treatment in Patients With Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Ipsen (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.101; HUM00151852 (Other: University of Michigan)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Nivolumab; irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nal-Irinotecan and Nivolumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: Nanoliposomal-Irinotecan; Drug: 5-Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Nivolumab — Intravenous (IV) infusion
  Other Names: Opdivo®, BMS-936558, MDX-1106, ONO-4538
Drug: Nanoliposomal-Irinotecan — Intravenous (IV) infusion
  Other Names: Onivyde®
Drug: 5-Fluorouracil — Intravenous (IV) infusion
  Other Names: 5-FU
Drug: Leucovorin — Intravenous (IV) infusion

SUMMARY:
The purpose of this study is to test the effectiveness (how well the drug works), safety, and tolerability of the investigational drug combination of nivolumab plus nanoliposomal-irinotecan, 5-fluorouracil, and leucovorin for patients with advanced or metastatic biliary tract cancer after progression on first-line systemic therapy.

ELIGIBILITY:
Inclusion

* Patients must have a pathologically confirmed carcinoma of the biliary tract (intra-hepatic, extra-hepatic (hilar, distal) or gall bladder) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors with mixed hepatocellular and cholangiocarcinoma histology are excluded.
* Patients must have received one and only one prior systemic therapy for advanced disease. Prior therapies must have not included irinotecan or PD- 1/PD-L1 antibody. Patient should have either progressed on or within 6 months of first-line systemic therapy or deemed intolerant of that therapy.
* Prior surgical resection, radiation, chemoembolization, radioembolization or other local ablative therapies are permitted if completed ≥ 4 weeks prior to registration AND if patient has recovered to ≤ grade 1 toxicity.
* Patients must have radiographically measurable disease (as per RECISTv1.1) in at least one site not previously treated with radiation or liver directed therapy (including bland, chemo- or radio-embolization, or ablation) either within the liver or in a metastatic lesion.
* Age ≥18 years
* Child-Pugh score of less than 7
* ECOG performance status of 0-1
* Ability to understand and willingness to sign IRB-approved informed consent
* Available archived tissue (FFPE block or 20 unstained slides from prior core biopsy or surgery)
* Must be able to tolerate CT and/or MRI with contrast
* Adequate organ function (per protocol) assessed ≤2 weeks prior to registration

Exclusion

* Must not have received systemic steroid therapy, or any other form of immunosuppressive therapy within 14 days prior to registration. Short bursts of steroids of 5-7 days (for COPD exacerbation or other similar indication) are allowed.
* No prior history of solid organ transplantation or brain metastasis (unless treated, asymptomatic and stable).
* Must not have undergone a major surgical procedure < 4 weeks prior to registration.
* Must not have an active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. Patients with history of malignancy are eligible provided primary treatment of that cancer was completed > 1 year prior to registration and the patient is free of clinical or radiologic evidence of recurrent or progressive malignancy.
* Must have no ongoing active, uncontrolled infections (afebrile for > 48 hours off antibiotics).
* Must not have received a live vaccine within 30 days of registration
* Must not have a psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.
* Women must not be pregnant or breastfeeding since 5-fluorouracil, nal- irinotecan and/or nivolumab may harm the fetus or child. All females of childbearing potential (not surgically sterilized and between menarche and 1- year post menopause) must have a blood test to rule out pregnancy within 2 weeks prior to registration.
* Women of child-bearing potential and men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation, and for 5 months (for women) and 7 months (for men) following completion of study therapy.
* Participants with an active, known or suspected autoimmune disease which may affect vital organ function, or has/may require systemic immunosuppressive therapy for management are excluded. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of registration are excluded. Inhaled, ocular, intra-articular, intra-nasal or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* No known UGT1A1* variants or Gilbert's syndrome
* Prisoners or subjects who are involuntarily incarcerated, or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness would be excluded.
* No known hypersensitivity to 5-fluorouracil, leucovorin, irinotecan, and/or nivolumab.
* Must not have ongoing bowel obstruction.
* No known HIV, Hepatitis B or Hepatitis C infection that is untreated and/or with a detectable viral load.
* Patients must not have uncontrolled intercurrent illness including, but not limited to, interstitial lung disease, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia.
* No known medical condition (e.g. a condition associated with uncontrolled diarrhea such as ulcerative colitis or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or interfere with the interpretation of safety results.
* Patients must not be on warfarin, strong CYP3A4 inducers (such as phenytoin, phenobarbital, primidone, carbamazepine, rifampin, rifabutin, rifapentine or St. John's wort), strong CYP3A4 inhibitors (such as ketoconazole, clarithromycin, indinavir, itraconazole, lopinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telaprevir, voriconazole), and strong UGT1A1 inhibitors (such as atazanavir, gemfibrozil, indinavir and ketoconazole).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Incidence of dose-limiting toxicities (DLTs) of drug combination nanoliposomal-Irinotecan, 5-fluorouracil, leucovorin and nivolumab | At 4 weeks after initiation of study treatment
  Adverse events will be graded according to NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0
Phase II: Median Progression-Free Survival (PFS) | Up to 2 years after last dose of study treatment or 3 years after first date of treatment initiation for those that remain on treatment
  Based on Kaplan-Meier estimates.

SECONDARY OUTCOMES:
Incidence of adverse events | Until discontinuation of study treatment, up to approximately 2 years after initiating study treatment or 3 years after first date of treatment initiation for those that remain on treatment
  Reportable adverse events are defined by the study protocol and graded according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) v5.0.
Overall Response Rate (ORR) | Up to 2 years after last dose of study treatment
  Determined per the combined Response Evaluation Criteria in Solid Tumours (RECISTv1.1) and immune-related RECIST (irRECIST) criteria
Median Overall Survival (OS) | Up to 2 years after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, MBBS, MS, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results published in peer reviewed research articles, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data is for meta-analysis, and has been approved by an independent review committee identified for this purpose. Proposals should be directed to vsahai@umich.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Sahai V, Griffith KA, Lin BS, Soares HP, Chandana SR, Crysler O, Kumar-Sinha C, Enzler T, Dippman D, Gunchick V, Zalupski MM. BilT03: Phase 1b/2 multicenter trial of nivolumab with 5-fluorouracil and liposomal irinotecan for previously treated advanced biliary tract cancer. Med. 2025 Apr 11;6(4):100547. doi: 10.1016/j.medj.2024.10.024. Epub 2024 Dec 18. PMID 39701097